CLINICAL TRIAL: NCT06627400
Title: Association of Urinary Incontinence With Depression, Insomnia, Frailty and Falls in Older Adults: a Cross-sectional Comprehensive Geriatric Assessment
Brief Title: Association of Urinary Incontinence With Depression, Insomnia, Frailty and Falls in Older Adults
Status: Completed | Type: Observational
Sponsor: Kastamonu University (Other)
Responsible Party: Principal Investigator, Sultan Keskin Demircan, Principal Investigator, Kastamonu University
Other Study IDs: Medical Doctor
Record Dates: First submitted 2024-09-30; First posted 2024-10-04 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Urinary Incontinence,Stress; Urinary Incontinence, Urge; Depressive Disorder; Insomnia; Frailty; Fall
MeSH Terms: conditions — Urinary Incontinence, Stress; Urinary Incontinence, Urge; Depressive Disorder; Sleep Initiation and Maintenance Disorders; Frailty

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 9 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of our study is to provide a holistic analysis of the geriatric syndromes associated with urinary incontinence, which can result in significant adverse outcomes in the elderly, and to explore the gender-specific relationships within these associations. The study revealed that urinary incontinence is highly prevalent among the older adults, particularly in women, and is associated strongly with depression, insomnia, frailty, and falls. Moreover, while older women with urinary incontinence exhibited more depressive symptoms than men, urinary incontinence was associated with similar frequencies of insomnia in both sexes. Considering the negative outcomes of depression, insomnia, frailty, and falls in older adults, as well as a decline in functionality, cognitive impairment, and prolonged hospitalizations and even mortality they cause, it becomes evident that urinary incontinence must be routinely assessed and treated by clinicians.

ELIGIBILITY:
Inclusion Criteria:

* The patients with comprehensive geriatric assessment data

Exclusion Criteria:

* dementia,
* those who experienced cerebrovascular occlusion with resulting neuromuscular paralysis
* active infections,
* schizoaffective disorder,
* epilepsy
* neuromuscular disorders
* those who were wheelchair or bed-bound,
* advanced chronic obstructive pulmonary disease (COPD)
* advanced chronic heart failure (CHF)

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study was conducted using the electronic records of patients aged 60 and over who presented to the outpatient geriatric clinic from January 2024 to July 2024. The patients with comprehensive geriatric assessment data were included in the study. Patients with dementia, those who experienced cerebrovascular occlusion with resulting neuromuscular paralysis, individuals with active infections, schizoaffective disorder, epilepsy or other neuromuscular disorders, as well as those who were wheelchair or bed-bound, and patients with advanced chronic obstructive pulmonary disease (COPD) and chronic heart failure (CHF) were excluded from the study.
Sampling Method: Probability Sample
Enrollment: 635 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-09-10 (Actual)

PRIMARY OUTCOMES:
depression | Baseline
  Yesavage Geriatric Depression Scale-short form;Scores above 4 were considered depression
frailty | Baseline
  Fried fraility index; Scores above 2 were considered frail
insomnia | Baseline
  The patient was asked if they had experienced complaints of insomnia in the last 1 months. if answer is yess, conisdered insomnia
fall history | Baseline
  The patient was asked if they had a history of falls in the past year.if answer is yess, conisdered fall history

CONTACTS AND LOCATIONS:
Locations (1):
- Kastamonu University, Kastamonu, Turkey (Türkiye)